CLINICAL TRIAL: NCT04331561
Title: Sensory Re-weighting Training for Orientation and Equilibrium: A Pilot Trial for the Treatment of Visually-induced Dizziness
Brief Title: Sensory Training for Orientation and Balance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0087; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 12/22/2020 (Other: UW Madison)
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Motion Sickness; Vertigo; Dizziness; Fall
MeSH Terms: conditions — Motion Sickness; Vertigo; Dizziness

STUDY DESIGN:
Intervention Model Description: Non-randomized, single group design with 2 baseline and 1 post-treatment assessment time points
Masking Description: Masking is not practical for this pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensory Re-weighting (Experimental): Adults with self-reported visually-induced dizziness will be recruited to help establish the feasibility and tolerability of the testing and training methods, as well as observe for any effects of the sensory re-weighting intervention. Tests involve assessing motion sickness, vision, somatosensation, balance, and perception of verticality. The treatment provided is designed to facilitate re-weighting of sensory feedback for orientation and balance. Participants will serve as their own controls.
  Interventions: Behavioral: sensory re-weighting

INTERVENTIONS:
Behavioral: sensory re-weighting — Participants will be supported in quiet standing by a safety harness and crisscrossing strap system. A cervical collar will be used to maintain consistent alignment between the head and trunk. A virtual reality headset is used to create a virtual environment in which visual stimuli will be presented. Three different body positions will be used during training: earth-vertical and clockwise and counterclockwise tilted 16º in the frontal plane. Sensory re-weighting will be driven by priming upregulation of somatosensory cues. In each training trial, participants must determine the direction of gravity and then indicate if the rod being displayed is aligned with gravity or if it needs to rotate clockwise or counterclockwise for that to be so. Participants will be instructed to pay attention to what they feel from their feet, legs, and gut during training and to use that pressure, stretch, movement, and muscle tension feedback to help them sense gravity.

SUMMARY:
This is a preliminary study of how human beings control balance and how symptoms of visually-induced dizziness may result in falls. The researchers created new tests of orientation and balance, as well as a new treatment for visually-induced dizziness. The researchers will use the new tests and treatments with adults who are affected by visually-induced dizziness. Testing is done twice before and once after treatment. The total time participants are involved in the study is approximately two weeks.

DETAILED DESCRIPTION:
This is a preliminary study of how human beings control balance and how symptoms of visually-induced dizziness may result in falls. The researchers created new tests of orientation and balance, as well as a new treatment for visually-induced dizziness. It is not known whether the new tests of orientation and balance are better, worse, or the same as existing tests in the ability to detect problems, nor is it known if the new treatment technique is any better, worse, or the same as existing treatments for dizziness and imbalance. However, the researchers hypothesize that the new tests will improve the ability to detect problems. They hypothesize that the treatment will result in less dizziness, better balance, and reduced risk of falling for those who receive it and that it is a better alternative to treatments that are already available to patients.

In order to see if this is true, the researchers will use the new tests and treatments with adults who are affected by dizziness. All participants in this study will undergo the same tests and will receive the same treatment. Testing is done twice before and once after the treatment period. The tests and treatment are done while standing on a computerized platform that measures balance and can tilt people from side to side. During these study procedures, participants wear virtual reality goggles that show them simple images in an otherwise dark environment.

The goal of the tests and the treatment is for participants to use what they feel to help them decide if the images shown inside the goggles are aligned with the person's sense of gravity. Participation in this study is voluntary and people who decide to participate may stop at any time without penalty.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have self-reported symptoms of visually-induced dizziness
* Participants must have normal self-reported cognitive function
* Participants must speak English fluently
* Weigh less than 225 pounds
* Be able to support their body weight in an upright posture for 15 minutes at a time
* Be able to follow the guidelines regarding permitted and prohibited additional treatments outlined in the study protocol.

Exclusion Criteria:

* Participants must not be participating in vestibular and balance rehabilitation therapy
* Pregnant or planning to become pregnant while in "on study" status
* Best-corrected visual acuity > 20/70
* Any self-reported, uncompensated, binocular vision abnormality, such as strabismus, amblyopia, or diplopia
* Peripheral neuropathy
* Self-reported history of frequent syncope (>1/month).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants Enrolled Relative to Approached | Up to 30 minutes
  Study feasibility is a primary outcome of this study. Feasibility will be measured using enrollment rates: the number of participants enrolled relative to the number of potential participants approached. This study will be considered 'feasible' with an enrollment rate higher than 70%
Participant Drop out Rate | Up to 3 weeks
  Tolerance of the intervention is a primary outcome of this study. Tolerance will be measured using the participant drop out rate. This study will be considered tolerable if the drop out rate is less than 20%
Post-Intervention Virtual Reality Sickness Questionnaire (VRSQ) Score | Visit 3 (Week 2)
  This questionnaire will be administered on paper immediately following each instance of testing and each round of training. Additional rest time will be required if participants symptoms are scored as > 33% on the VRSQ (see below for more information regarding VRSQ scoring). Symptoms must return to baseline before participants are permitted to begin a round of testing or training. The VRSQ is comprised of nine items from two domains (oculomotor: general discomfort, fatigue, eye strain, and difficulty focusing; disorientation: headache, fullness of head, blurred vision, dizzy (eyes closed), and vertigo). The intensity of each item is rated on a 4-point Likert scale: 0 = not at all, 1 = slightly, 2 = moderately, and 3 = very. Scores for each sub-scale and the total score range from 0 to 100. Higher scores indicate greater symptom intensity. The VRSQ is an adaptation of the Simulator Sickness Questionnaire (SSQ) for use in virtual environments.

SECONDARY OUTCOMES:
Change in Motion Sensitivity Assessment Questionnaire (MSAQ) Overall Score | Visit 1 (Week 1) and Visit 3 (Week 2)
  The MSAQ was designed to evaluate symptoms of visually-induced motion sickness in response to an optokinetic stimulus. Respondents use a 9-point scale to indicate how accurately 16 statements describe their experience viewing the stimulus. Statements include, "I felt sick to my stomach" and "I felt dizzy." The overall score is obtained by calculating the percentage of total points scored: (sum of points from all items/144) × 100. Higher scores indicate greater severity of symptoms. The MSAQ will be administered on paper following exposure to an optokinetic stimulus while standing and wearing the virtual reality headset. Participants will rate their symptoms on the MSAQ after 1 minute of exposure to an annulus rotating clockwise and counterclockwise at 30 degrees per second. Participants will be permitted to rest with the headset off between the clockwise and counterclockwise trials until symptoms have completely resolved. The reliability and validity of the MSAQ have been established.
Change in Visual Vertical Analogue Scale (VVAS) Total Score | Visit 1 (Week 1), Visit 2 (in Week 2), Visit 3 (in Week 2)
  The VVAS consists of nine scales, each relating to a specific symptom-provoking situation. A revision of the VVAS by researchers at the University of Pittsburgh is in press. The revised version consists of 15 scales. The revised version will be administered in this study. In the revised version of the VVAS, each scale has two anchors, 0 representing no dizziness and 10 representing extreme dizziness or activity avoidance. The distance from the zero anchor to the respondent's marking is measured electronically. Items that are not applicable to the individual's life may be completed as imagined. Internal consistency and validity of the VVAS have been established. A total score is calculated to determine the severity of visual vertigo by summing all items, dividing by the number of answered items, and then multiplying by 10. The maximum score is 100 with higher scores indicating greater symptom severity.
Change in Vision-related Dizziness Questionnaire (VRDQ) Total Score | Visit 1 (Week 1), Visit 2 (in Week 2), Visit 3 (in Week 2)
  The VRDQ is used to quantify vision-related dizziness. This outcome measure consists of 25 questions comprising two subscales [frequency and severity of symptoms]. The maximum score for each sub-scale is 100 points. The total score is the average of both sub-scales. Higher scores represent greater frequency and severity of symptoms. Test-retest reliability for the VRDQ is well above the good performance level and convergent validity for the VRDQ was demonstrated with the Dizziness Handicap Inventory (DHI). Spearman correlation coefficients are 0.75 between the DHI and VRDQ frequency scale and 0.76 between the DHI and VRDQ severity scale.
Change in Rod and Disk Test (RDT) Mean Performance | Visit 1 (Week 1), Visit 2 (in Week 2), Visit 3 (in Week 2)
  The image of an annulus comprised of a pseudorandomized pattern of dots will be presented in the virtual reality headset. The image of a rod is also presented within the central region of the annulus that is black. This image will be rotated at 30° per second in either a clockwise or counterclockwise direction around the participant's line of sight. A batch of rod angles will be predetermined. This assessment will be completed using an Oculus Rift and without reference to external visual cues. Only binocular testing will be completed. The average value for performance in each position will be used in data analysis. The mean of absolute value of the error in rod alignment measured in degrees for each body position tested will be used as the measurement variable for this outcome. Mean performance in this population is 15.1 (sd 8.4). Higher values indicate greater deviation of perceived vertical from earth vertical.
Change in Subjective Visual Vertical (SVV) Mean Performance | Visit 1 (Week 1), Visit 2 (in Week 2), Visit 3 (in Week 2)
  An image of a rod will be shown in the central portion of the visual field. The surrounding virtual environment will be void. A batch of rod angles will be predetermined. This assessment will be completed using an Oculus Rift and without any reference to external visual cues. Only binocular testing will be completed. The average value for performance in each position will be used in data analysis. The mean of absolute value of the error in rod alignment measured in degrees for each body position tested will be used as the measurement variable for this outcome. Mean performance in this population is 0.39 (sd 0.8). Higher scores indicate subjective visual vertical alignment that is farther away from earth vertical.
Change in Rod and Frame Test (RFT) Mean Performance | Visit 1 (Week 1), Visit 2 (in Week 2), Visit 3 (in Week 2)
  An image of a rod will be projected inside a tilted frame within the central portion of the visual field. The surrounding virtual environment will be void. The frame will be tilted by +/- 20° in the frontal plane. A batch of rod angles will be predetermined. This assessment will be completed using an Oculus Rift and without reference to external visual cues. Only binocular testing will be completed. The average value for performance in each position will be used in data analysis. The mean of absolute value of the error in rod alignment measured in degrees for each body position tested will be used as the measurement variable for this outcome. Mean performance in this population is 6.51 (sd 7.8). Higher values indicate greater deviations of perceived vertical from earth vertical.
Change in Multisensory Balance Evaluation (MBE) as measured by the Intersection Point Height | Visit 1 (Week 1), Visit 2 (in Week 2), Visit 3 (in Week 2)
  This test is designed to assess balance during quiet standing in different sensory conditions. Participants perform one trial (lasting 50 seconds) of each condition. All trials are performed while standing on a force plate with the feet in a self-selected, comfortable position. The force plate samples center of pressure and direction of ground reaction force. The visual environment is controlled using an Oculus Rift. The surface conditions are either non-compliant or compliant. The frequency-dependent height of the Intersection Point (IP) of the ground reaction force is the main outcome. The behavior and shape of the IP curvature will be studied in each test trial. The IP curvature for certain conditions will be compared versus others in order to assess the impact of manipulating specific sensory inputs on the behavior of the IP. The height of the IP at a specific frequency represents how stable a person is during a given test trial. Lower IP height suggests greater stability.
Change in Semmes-Weinstein Monofilament Examination (SWME) Discrimination Threshold | Visit 2 (in Week 2) and Visit 3 (in Week 2)
  A SWME will be conducted at the pre-test 2 and post-test 1 assessments in order to determine if the sensory re-weighting training results in changes in sensitivity to light touch/deep pressure sensation on the soles of the feet. Lower SWME threshold indicate increased sensitivity to light touch. The sensitivity between 0.008 grams and 2.0 grams will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kreg G Gruben, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
The research team does not plan to share individual participant data.